CLINICAL TRIAL: NCT03905915
Title: The Impact of Induced Hypnosis by Virtual Reality AQUA Module on Preoperative Anxiety.
Brief Title: Virtual Reality (VR) to Reduce Preoperative Anxiety.
Acronym: RVAQUA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Roelants, Clinical professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/20JUL/345
Record Dates: First submitted 2019-03-26; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Preoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative virtual reality session (Other): Amsterdam Anxiety score recorded before VR session is followed by a 15 min VR session and finally Amsterdam Anxiety score is recorded after VR session
  Interventions: Device: Virtual reality (VR) session with AQUA module

INTERVENTIONS:
Device: Virtual reality (VR) session with AQUA module — A device with virtual reality is given to the patients with a film of 15 minutes

SUMMARY:
Most patients awaiting surgery show significant anxiety score which can be influenced by the fear of anesthesia or surgery but also by the context of care. These anxious patients will have more postoperative complications and can also develop chronic pain. The Virtual reality AQUA module induces hypnosis and is specially designed to reduce anxiety. The purpose of the study is to examine the effect of a virtual reality session on preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing scheduled orthopedic surgery with loco-regional anesthesia at Saint-Luc Hospital.
* Patients not following long-term psychotherapeutic treatment
* Patients not taking psychotropic medication
* free, informed and written consent signed by the investigator and the patient before the procedure.

Exclusion Criteria:

* patient not speaking French
* Patients with long-term psychotherapeutic treatment
* Patients taking psychotropic drugs
* patient blind and deaf

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Amsterdam preoperative anxiety and information score (APAIS) after VR session | 5 minutes after virtual reality session
  The Amsterdam preoperative anxiety and information (APAIS) scale is a 6-items questionnaire. Each item is scored from 1(not at all) to 5(extremely). 4 items assess anxiety (patient with a score >or = to 11 is considered very anxious), 2 items assess the desire for information (patient with a score > 8 is considered very anxious because there is a corelation between need for informa tion and anxiety). The score ranges from 6 (no anxious) to 30 (highly anxious).

SECONDARY OUTCOMES:
Evaluation du Vécu de l'ANesthésie - LocoRégionale) EVAN-LR satisfaction score | 2 hours after VR session (in the recovery room, after surgery)
  Evaluation du Vécu de l'Anesthésie LocoRégionale (EVAN-LR) is a tool assessing patient satisfaction within the perioperative period surrounding regional anesthesia. The EVAN-LR comprises 19 items, structured in a global index and five dimensions: Attention, Information, Discomfort, Waiting, and Pain. Each item is scored from 1(not at all) to 5(extremely). The score ranges from 18(no satisfied) to 95 (highly satisfied).
Change of Visual Analog Score (VAS) anxiety score after VR session | 5 minutes after the virtual reality session
  score between 0 ( no anxious) and 10 (highly anxious)

CONTACTS AND LOCATIONS:
Overall Officials: Roelants Fabienne, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruhaiyem ME, Alshehri AA, Saade M, Shoabi TA, Zahoor H, Tawfeeq NA. Fear of going under general anesthesia: A cross-sectional study. Saudi J Anaesth. 2016 Jul-Sep;10(3):317-21. doi: 10.4103/1658-354X.179094. PMID 27375388
- [Result] Scavee V, Dehullu JP, Scavee JP, Michel I. Impact of Anxiety in Ambulatory Superficial Venous Surgery : A Prospective Study Using the HADS-A Scale. Acta Chir Belg. 2015 Jan-Feb;115:42-8. PMID 26021790
- [Result] Ganry L, Hersant B, Sidahmed-Mezi M, Dhonneur G, Meningaud JP. Using virtual reality to control preoperative anxiety in ambulatory surgery patients: A pilot study in maxillofacial and plastic surgery. J Stomatol Oral Maxillofac Surg. 2018 Sep;119(4):257-261. doi: 10.1016/j.jormas.2017.12.010. Epub 2018 Jan 6. PMID 29317347
- [Result] Maurice-Szamburski A, Bruder N, Loundou A, Capdevila X, Auquier P. Development and validation of a perioperative satisfaction questionnaire in regional anesthesia. Anesthesiology. 2013 Jan;118(1):78-87. doi: 10.1097/ALN.0b013e31827469f2. PMID 23221859
- [Result] Maurice-Szamburski A, Loundou A, Capdevila X, Bruder N, Auquier P. Validation of the French version of the Amsterdam preoperative anxiety and information scale (APAIS). Health Qual Life Outcomes. 2013 Oct 7;11:166. doi: 10.1186/1477-7525-11-166. PMID 24099176